CLINICAL TRIAL: NCT03774602
Title: Evaluation of the Maternal and Child Survival Program (MCSP) in Mozambique Using Mixed Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jhpiego (Other)
Collaborators: Ministry of Health, Mozambique (Other Government); United States Agency for International Development (USAID) (U.S. Federal Agency); Save the Children (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB 8902
Record Dates: First submitted 2018-12-11; First posted 2018-12-13 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Knowledge, Attitudes, Practice; Gender Issues
MeSH Terms: conditions — Behavior; Sexism | interventions — Health Promotion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MCSP package of interventions (Experimental): MCSP package of interventions for health promotion and provision of RMNCH services
  Interventions: Behavioral: Health promotion and provision of RMNCH services

INTERVENTIONS:
Behavioral: Health promotion and provision of RMNCH services — Implementation of quality, high-impact interventions at institutional and community levels to increase access to and utilization of RMNCH services

SUMMARY:
This study evaluates changes in knowledge, attitudes, practices and coverage of key reproductive, maternal, newborn, and child health (RMNCH) areas, including malaria, family planning (FP), nutrition, water, sanitation and hygiene (WASH), and gender equity among the population in Nampula and Sofala provinces targeted by the Maternal and Child Survival Program (MCSP) in Mozambique.

DETAILED DESCRIPTION:
The specific objectives of the study are to:

1. Assess changes in knowledge, attitudes, practices and coverage (KAPC) of high-impact interventions related to MNCH (antenatal care, delivery, post-partum/natal care, and sick child care), immunization, family planning and reproductive health, nutrition, WASH and malaria among mothers and fathers of children age 0-23 months in MCSP supported areas;
2. Evaluate the effectiveness of male engagement interventions that encourage couples communication at increasing antenatal care (ANC) attendance, joint birth preparedness and complication readiness (BPCR) plans, institutional birth, and use of modern FP;
3. Determine the feasibility and acceptability of male engagement interventions on RMNCH services for clients and providers;
4. Explore how decisions between couples are made and what may influence their decisions about seeking RMNCH services; and
5. Explore the experiences of women who were referred to a health facility for themselves or their child for obstetric, newborn or child health complications, and examine the factors contributing to whether and how those referrals were completed in Nampula Province.

This study is a final program evaluation that will use a mixed methods approach, including both quantitative and qualitative data collection.

Quantitative data will be collected through a cross-sectional KAPC household survey of mothers and fathers of children age 0-23 months, replicating the same KAPC questionnaire that was conducted at baseline in 2016 in the same geographic areas. Questions were harmonized with the DHS and MICS where appropriate. Findings from the endline KAPC survey will be compared to findings from the baseline survey to assess changes over time in the primary outcomes of interest.

Qualitative data will be collected through focus group discussions (FGDs) and in-depth interviews (IDIs) with clients (mothers and fathers of children age 0-23 months) and health providers in MCSP-supported areas. The qualitative component will be conducted to help us gain a more in-depth understanding of the influence of male engagement interventions on couples' decision-making and care-seeking related to RMNCH as well as the barriers and facilitators that affected the experience of identified women who were referred to health facilities for obstetric or newborn complications. We will explore both client and provider experiences with gender-equitable male engagement practices, as well as individual client referral narratives related to obstetric or newborn complications.

ELIGIBILITY:
Inclusion Criteria (KAPC survey):

* Women 15 years and older who have had a live birth in the 2 years preceding the survey and the child is living at the time of the interview
* Male partners (age 18 and older) of women 15 years and older who have had a live birth in the 2 years preceding the survey and the child is living at the time of the interview

Exclusion Criteria (KAPC survey): Women 15-17 years without parent permission to participate in study

Inclusion Criteria (Referral narrative interviews): Women who: a) delivered in the last 12 months who experienced obstetric complications; b) whose newborn experienced complications in the last year; c) whose child 0-59 months experienced an illness in the last year

Inclusion Criteria (Provider interviews):

* Facility managers working in selected primary health care centers
* Health care workers who provide RMNCH services in MCSP-supported facility in one of these six areas: ANC, maternity, postnatal care, FP, sick child, or well-child

Exclusion Criteria (Provider interviews): Has been working in the facility for < 6 months

Inclusion Criteria (Male engagement FGDs):

* Women 18-49 years of age who delivered in the last 12 months
* Male partner (age 18 and older) of a woman 18-49 years of age who delivered in the last 12 months
* Participated in a community dialogue

Ages: 15 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2767 (Actual)
Dates: Start 2018-11-22 (Actual); Primary Completion 2018-12-22 (Actual); Study Completion 2018-12-22 (Actual)

PRIMARY OUTCOMES:
Institutional delivery rate | 2 years
  Percentage of last-born children age 0-23 months who were born in a health facility
Percentage of pregnant women who had four or more ANC visits | 2 years
  Percentage of mothers of children age 0-23 months who had four or more antenatal care visits while pregnant with their youngest child
Percentage of children under 2 years of age who received Penta 1 vaccination but did not receive Penta 3 (Drop out rate) | 2 years
  Percentage of children age 12-23 months who received a Penta 1 vaccination but did not receive a Penta 3 vaccination according to or card verified at the time of the survey
Percentage of mothers who made birth preparations before giving birth | 2 years
  Percentage of mothers of children age 0-23 months who made birth preparations before the birth of their youngest child

SECONDARY OUTCOMES:
Percentage of women who have discussed FP use with her partner | 2 years
  Percentage of women of reproductive age who have discussed with her partner whether to use a FP method
Percent of infants under 6 months of age who are exclusively breastfed | 2 years
  Percentage of infants 0-5 months of age who are fed exclusively with breast milk

CONTACTS AND LOCATIONS:
Overall Officials: Connie Lee, MPH, MIA, Principal Investigator — Jhpiego
Locations (21):
- Mozambique (21):
  - Angoche District, Community Setting, Angoche, Nampula
  - Meconta District, Community Setting, Meconta, Nampula
  - Mecuburi District, Community Setting, Mecubúri, Nampula
  - Moma District, Community Setting, Moma, Nampula
  - Monapo District, Community Setting, Monapo, Nampula
  - Mossuril District, Community Setting, Mossuril, Nampula
  - Centro de Saude Ontupaia, Nacala, Nampula
  - Centro de Saude Quissinmanjulo, Nacala, Nampula
  - Nacala Porto District, Community Setting, Nacala, Nampula
  - Erati District, Community Setting, Namapa-erati, Nampula
  - Centro de Saude Iapala Sede, Ribáuè, Nampula
  - Hospital Rural de Ribaue, Ribáuè, Nampula
  - Ribaue District, Community Setting, Ribáuè, Nampula
  - Beira City, Community Setting, Beira, Sofala
  - Buzi District, Community Setting, Búzi, Sofala
  - Centro de Saude Ampara, Búzi, Sofala
  - Centro de Saude Bandua, Búzi, Sofala
  - Dondo District, Community Setting, Dondo, Sofala
  - Centro de Saude Metuchira, Nhamatanda, Sofala
  - Hospital Rural de Nhamatanda, Nhamatanda, Sofala
  - Nhamatanda District, Community Setting, Nhamatanda, Sofala

IPD SHARING:
Plan to Share IPD: Undecided